CLINICAL TRIAL: NCT00855530
Title: A Fifty-Two-Week Multicenter, Open-Label, Study Evaluating the Long-Term Safety and Tolerability of SR58611A 350 mg q12 in Patients With Major Depressive Disorder.
Brief Title: Long Term Safety and Tolerability of SR58611 in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS4848
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Major Depressive Disorders
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — amibegron; Amibegron hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: amibegron (SR58611A)

INTERVENTIONS:
Drug: amibegron (SR58611A) — oral administration of 300 mg twice daily

SUMMARY:
Primary objective:

- To evaluate the long-term safety and tolerability of SR58611A (amibegron) patients with major depressive disorder (MDD).

Secondary objective:

- To determine plasma concentrations of SR58878 (the active metabolite of SR58611A), for pharmacokinetic population analyses, to evaluate the quality of life (QoL) in patients with MDD, and to evaluate the efficacy of amibegron in patients with MDD.

ELIGIBILITY:
Inclusion Criteria:

* patients as defined by Diagnosis and Statistical Manual of Mental Disorders, recurrent episode for at least 1 month prior to entry into the study, and with a total score of > 18 on the Hamilton Depression Rating Scale (HAM-D) 17-items.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2005-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Clinical monitoring of adverse events (AEs), laboratory parameters, vital signs, physical examinations, and physician withdrawal checklists | 54 weeks

SECONDARY OUTCOMES:
17-item Hamilton Depression rating Scale, Clinical Global Impression, Sheehan Disability Scale, Qol Enjoyment and satisfaction Questionnaire - Short Form,Medical Outcomes Study Short Form, Endicott Work Productivity Scale. | 54 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (11):
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Causeway Bay, Hong Kong
- Sanofi-Aventis Administrative Office, Casablanca, Morocco
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Mégrine, Tunisia